CLINICAL TRIAL: NCT01919047
Title: Drug Use-Results Survey of Betanis Tablets 25 and 50 mg
Brief Title: Drug Use-Results Survey of Betanis Tablets in Japan
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: BE0001
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; mirabegron; occurrence of adverse events; Overactive Bladder Symptom Score
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Betanis group: Patients receiving Betanis for Overactive Bladder
  Interventions: Drug: Betanis

INTERVENTIONS:
Drug: Betanis — Oral
  Other Names: Mirabegron; YM178

SUMMARY:
This study is to determine the following information.

1. The occurrence of adverse drug reactions in clinical settings.
2. Factors potentially impacting safety, effectiveness, and other aspects.

DETAILED DESCRIPTION:
This survey aims to determine the following information and the need for conducting specified drug use-results surveys and post-marketing clinical studies in patients using Betanis (generic name: mirabegron):

1. The occurrence of adverse drug reactions in clinical settings.
2. Factors potentially impacting safety, effectiveness, and other aspects.

Items of Particular Interest:

* Safety and effectiveness in patients with hepatic impairment and patients with renal impairment.
* Safety and effectiveness when mirabegron is used concomitantly with other drugs (α1 blockers, anticholinergic agents, 5α reductase inhibitors, drugs with a potent CYP3A4-inhibiting effect, drugs with a CYP3A4-inducing effect, drugs metabolized primarily by CYP2D6, and other frequently used drugs).
* The occurrence of cardiovascular adverse events.
* The occurrence of adverse events related to increased intraocular pressure.
* The occurrence of urinary retention

ELIGIBILITY:
Inclusion Criteria:

* Patients who received mirabegron for the first time for the treatment of urinary urgency, daytime frequency, and urgency incontinence associated with overactive bladder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received mirabegron for the first time for the treatment of urinary urgency, daytime frequency, and urgency incontinence associated with overactive bladder.
Sampling Method: Non-Probability Sample
Enrollment: 10711 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and adverse drug reactions | For 12 weeks

SECONDARY OUTCOMES:
Changes in OABSS (overactive bladder symptom score) | baseline and at 12 weeks (or last observation period)
Items of particular interest | baseline and at 12 weeks (or last observation period)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku